CLINICAL TRIAL: NCT06061679
Title: Impact of Switching COPD Patients From Inhaler Devices to the Omron C28P Nebuliser: a Prospective, Real-world Study
Brief Title: Impact of Switching COPD Patients From Inhaler Devices to the Omron C28P Nebuliser.
Acronym: OMRON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University of Florence, UNIFI University of Florence, Florence, Italy Florence (Unknown)
Responsible Party: Principal Investigator, BONINI MATTEO, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5432
Record Dates: First submitted 2023-09-01; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease) With Acute Lower Respiratory Infection
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Open, single-arm, real-life, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omron C28P cohort (Experimental): Patients diagnosed with COPD using the study device (OMRONC28P) for 24 weeks.
  Interventions: Device: Omron C28P nebuliser

INTERVENTIONS:
Device: Omron C28P nebuliser — switch from portable inhalers to the Omron C28P nebuliser

SUMMARY:
The cornerstone of COPD therapy is based on the use of inhalation drugs. The correct use of devices is crucial; a suboptimal use technique is the cause of a possible clinical deterioration with a consequent increase in exacerbations and healthcare expenditure. Inhalation of drugs by nebulizer, in specific populations of patients who have shown poor adherence to inhalation therapy and poor symptomatological control, could be a more advantageous therapeutic strategy than pMDIs or DPIs, not requiring coordination at the time of delivery and not requiring an effective inspiratory effort.

The objective of this study is to evaluate the effects of the transition from portable inhalers (pMDIs or DPIs) to an innovative prototype Omron C28P nebulizer, measured primarily as changes in treatment adhesion and respiratory symptoms. The sudy design is open, single-arm, real-life, prospective study conducted in two tertiary level respiratory centers in Italy, with assessments conducted on the occasion of patients' visits to their doctor.

DETAILED DESCRIPTION:
The cornerstone of pharmacological treatment of COPD is represented by bronchodilator and corticosteroid medications delivered by pressurised metered-dose inhalers (pMDIs) and dry powder inhalers (DPIs). Any inhaler device category can be equally effective in treating patients if properly used. However, each device exhibits distinct properties that warrant consideration in achieving successful medication delivery. Errors frequently observed in patients with obstructive pulmonary diseases are incorrect coordination between inspiration and pMDIs activation and insufficient inspiratory effort or wrong device preparation with DPIs. Suboptimal inhaler technique is the prominent reason for the lack of efficacy and can contribute to poor adherence to medications that, in turn, is associated with worsening in disease control, increased rate of exacerbations, increased healthcare resource consumption, and consequently increased healthcare expenditure. Inhaler devices, which may seem simple to use to healthcare providers, frequently present challenges particularly for elderly patients with COPD. The combined effects of co-morbidities, the complexity of the accompanying medication regimens, as well as age- and disease-related lung function decline may add to the complexity of using different inhalers.

Once set up, nebulisers are easier for patients to use than pMDIs or DPIs as they only require tidal respiration for effective drug delivery with, therefore, no need to coordinate inspiration with device activation as for pMDIs, or to require high inspiratory effort as for DPIs. The primary aim of the present study is to assess the effect on inhaler adherence and disease control of switching patients from their portable inhalers (either pMDIs or DPIs) to the Omron C28P nebuliser, as assessed by means of the Test of Adherence to Inhalers (TAI) questionnaire and the COPD Assessment Test (CAT), respectively. The investigators plan to enroll 99 adult outpatients of both genders with a diagnosis of COPD of any functional severity; a sample size of 99 patients was chosen to design the study to have a 80% statistical power of detecting a difference of 2.07 (±1.03 SD) and of 3 (±5 SD) in TAI and CAT score, respectively, after device switching. The study consists of a baseline (T0) and 2 follow-up visits at 8 (T1) and 24 (T2) weeks (±2) after enrolment. On each study visit, after completion of clinical history and measurements of vital parameters, patients will be requested to rate their adherence to inhalers by filling the TAI questionnaire. Impact of COPD on health status and dyspnoea perception will be assessed by measuring the CAT score and the mMRC score. After completion of the above-mentioned procedures, patients will be carefully instructed by trained investigators on the use of the Omron C28P nebuliser. To this end, practical session with the nebuliser and dedicated videos will be used.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients treated by inhaled bronchodilators, corticosteroids or their combinations delivered by inhaler devices
* COPD patients not adherent (TAI ≤ 45) to recommended therapy
* COPD patients with a CAT score ≥18.
* Must be capable of giving informed consent to participate, and available to comply with the requirements and procedures foreseen by the study protocol.

Exclusion Criteria:

* COPD patients with history of recent (< 4 weeks) upper respiratory tract infections and/or airways exacerbations
* patients with recent (< 2 months) pulmonary surgery or any active diseases that, in the judgement of the investigator, may interfere with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The primary aim of the present study is to assess the effect on inhaler adherence to the Omron C28P | 24 weeks
  The primary aim of the present study is to assess the effect on inhaler adherence to the Omron C28P, assessed by means of the Test of Adherence to Inhalers (TAI) questionnaire
The co-primary aim of the present study is to assess the effect on disease control of switching patients from their portable inhalers (either pMDIs or DPIs) to the Omron C28P | 24 weeks
  The co-primary aim of the present study is to assess the effect on disease control of switching patients from their portable inhalers (either pMDIs or DPIs) to the Omron C28P assessed by means of the COPD Assessment Test (CAT)